CLINICAL TRIAL: NCT00741429
Title: A 2-Month Safety Follow-up Trial of Subjects From MannKind Protocols MKC-TI-009, MKC-TI-102, MKC-TI-103 and MKC-TI-030
Brief Title: A 2-Month Safety Follow-Up Trial
Status: Completed | Type: Observational
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MKC-TI-126
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Ex-TI: Ex-Technosphere® Insulin Inhalation Powder (subjects previously received TI Inhalation Powder)
  Interventions: Drug: Technosphere Insulin Inhalation Powder
- Non Ex-TI: Non Ex-Technosphere® Insulin Inhalation Powder (subjects previously received another anti-diabetic medication)
  Interventions: Drug: Comparator

INTERVENTIONS:
Drug: Technosphere Insulin Inhalation Powder — Subjects previously treated with Technosphere Insulin Inhalation Powder
  Groups: Ex-TI
Drug: Comparator — Subjects previously treated with other anti-diabetic medications
  Groups: Non Ex-TI

SUMMARY:
The main purpose of the trial is to evaluate pulmonary function in subjects who had completed any one of the 4 MKC parent trials (MKC-TI-009, MKC-TI-102, MKC-TI-103, or MKC-TI-030) for an additional 2-month safety follow-up.

DETAILED DESCRIPTION:
This was a 2-month safety follow-up study of subjects from MannKind protocols MKC-TI-009, MKC-TI-102, MKC-TI-103 and MKC-TI-030. No study medications were administered during this trial. The adverse event data included are for the combined Safety population irrespective of previous treatments in the parent trials.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed any of the 4 MKC parent trials (MKC-TI-103, MKC-TI-009, MKC-TI-102, MKC-TI-030)
* Urine cotinine test of less than or equal to 100 ng/mL
* Written informed consent

Exclusion Criteria:

* Subjects who started smoking during the 4 week follow-up phase of the parent trial
* Subjects who began a new inhaled insulin regimen with an investigational drug during the 4 week follow-up phase of the parent trial and/or are participation in another clinical trial
* Female subjects who are pregnant, lactating or planning on becoming pregnant
* Subjects with a positive urine drug screening at Visit 1
* Female subjects of child-bearing potential not practicing adequate birth control

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of eligible type 1 and type 2 diabetic subjects who have completed any of the 4 MKC parent trials (MKC-TI-103, MKC-TI-009, MKC-TI-102, MKC-TI-030).
Sampling Method: Non-Probability Sample
Enrollment: 649 (Actual)
Dates: Start 2007-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 (L) from Baseline Visit in Parent Trial to Visit 2 of MKC-TI-126 | 9 to 27 months

SECONDARY OUTCOMES:
Change in FVC (L) from Baseline Visit in Parent Trial to Visit 2 of MKC-TI-126 | 9 to 27 months
Change in TLC (L) from Baseline Visit in Parent Trial to Visit 2 of MKC-TI-126 | 9 to 27 months
Change in Hemoglobin Corrected DLco (mL/min/mm Hg) from Baseline Visit in Parent Trial to Visit 2 of MKC-TI-126 | 9 to 27 months
Change in FEV1 (L) from Final Assessment of Treatment Phase in Parent Trial to Visit 2 of MKC-TI-126 | 3 Months
Change in FVC (L) from Final Assessment of Treatment Phase in Parent Trial to Visit 2 of MKC-TI-126 | 3 Months
Change in TLC (L) from Final Assessment of Treatment Phase in Parent Trial to Visit 2 of MKC-TI-126 | 3 Months
Change in Hemoglobin Corrected DLco (mL/min/mmHg) from Final Assessment of Treatment Phase in Parent Trial to Visit 2 of MKC-TI-126 | 3 Months

CONTACTS AND LOCATIONS:
Locations (150):
- United States (109):
  - Parkway Medical Center, Birmingham, Alabama
  - Coastal Clinical Research Inc, Mobile, Alabama
  - Radiant Research (Phoenix), Chandler, Arizona
  - Southwest Health Ltd Research Division, Phoenix, Arizona
  - Northwest Medical Center, Phoenix, Arizona
  - Canyon Clinical Research, Tucson, Arizona
  - Arizona Research Associates, Tuscon, Arizona
  - Private Practice, Burlingame, California
  - International Clinical Research Network, Chula Vista, California
  - Family Medical Center, Foothill Ranch, California
  - Saad Hijazi MD Inc, Fresno, California
  - Saint Agnes Medical Center, Fresno, California
  - Valley Research, Fresno, California
  - Digestive & Liver Disease Specialist A Medical Group Inc, Garden Grove, California
  - Diabetes/Lipid Management and Research Center, Huntington Beach, California
  - Interlink Research Institute, Los Alamitos, California
  - Southern California Endocrine Center, Pasadena, California
  - Dorothy L & James E Frank Diabetes Research Institute, San Mateo, California
  - Sansum Medical Research Institute, Santa Barbara, California
  - Coastal Biomedical Research Inc, Santa Monica, California
  - Encompass Clinical Research, Spring Valley, California
  - Diabetes Research Center, Tustin, California
  - Creekside Endocrine Associates, Denver, Colorado
  - Chase Medical Research LLC, Waterbury, Connecticut
  - Center for Diabetes & Endocrine Care, Hollywood, Florida
  - University of Miami Diabetes Research Institute, Miami, Florida
  - International Research Associates LLC, Miami, Florida
  - Laureate Clinical Research Group, Atlanta, Georgia
  - Executive Health and Research Associates Inc, Atlanta, Georgia
  - Rockdale Medical Research Associates, Conyers, Georgia
  - Private Practice, Decatur, Georgia
  - Atlanta Pharmaceutical Research Center, Dunwoody, Georgia
  - North Atlanta Endocrinology & Diabetes PC, Lawrenceville, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Cedar-Crosse Research Center, Chicago, Illinois
  - John H Stoger Jr Hospital of Cook County, Chicago, Illinois
  - MODEL Clinical Research, Baltimore, Maryland
  - Health Trends Research LLC, Baltimore, Maryland
  - Franklin Square Hospital, Baltimore, Maryland
  - James A Dicke MDPA, Towson, Maryland
  - Hurley Medical Center, Flint, Michigan
  - KMED Research, Saint Clair Shores, Michigan
  - Radiant Research Inc (Minneapolis), Edina, Minnesota
  - Center for Urologic Clinical Trials University of Minnesota, Minneapolis, Minnesota
  - Amin Radparvar's Private Practice, City of Saint Peters, Missouri
  - Healthcare Research, Florissant, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Clayton Medical Research, St Louis, Missouri
  - MedEx Healthcare Research Inc(009), St Louis, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Deaconess Billings Clinic Research Center, Billings, Montana
  - Montana Health Research Institute, Billings, Montana
  - Creighton Diabetes Center, Omaha, Nebraska
  - Your Doctors Care, Hillsborough, New Jersey
  - Hopewell Valley Medical Group, Trenton, New Jersey
  - Umdnj-Som, Voorhees Township, New Jersey
  - New Mexico Clinical Research & Osteoporosis Center, Albuquerque, New Mexico
  - Lovelace Scientific Resources (Albuquerque), Albuquerque, New Mexico
  - Southwest Endocrinology Associates, Albuquerque, New Mexico
  - University of New Mexico HCS, Albuquerque, New Mexico
  - Diabetes Care & Information Center of New York, Flushing, New York
  - Winthrop University Hospital, Mineola, New York
  - North Shore Diabetes and Endocrine Associates, New Hyde Park, New York
  - M.E.R.I., New York, New York
  - Univeristy of Physicians Group Endocrine Division, Staten Island, New York
  - Metrolina Medical Research, Charlotte, North Carolina
  - Sensenbrenner Primary Care, Charlotte, North Carolina
  - Physician's East PA, Greenville, North Carolina
  - Rapid Medical Research Inc, Cleveland, Ohio
  - Providence Health Partners - Center of Clinical Research, Dayton, Ohio
  - Wells Institute for Health Awareness, Kettering, Ohio
  - Your Diabetes Endocrine Nutrition Group, Mentor, Ohio
  - Portland Diabetes & Endocrinology Center, Portland, Oregon
  - Legacy Clinical Research, Portland, Oregon
  - Covance CRU Inc., Portland, Oregon
  - Bucks County Clinical Research, Morrisville, Pennsylvania
  - Upstate Pharmaceutical Research, Greenville, South Carolina
  - Southeastern Research Associates Inc, Taylors, South Carolina
  - AM Diabetes and Endocrinology Center, Bartlett, Tennessee
  - Collierville Medical Specialists, Collierville, Tennessee
  - Memphis Internal Medicine PLLC, Memphis, Tennessee
  - Israel Hartman MD, Arlington, Texas
  - Texas Familicare Clinical Research, Colleyville, Texas
  - Dallas Diabetes & Endocrine Center, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Radiant Research Dallas-North, Dallas, Texas
  - Baylor Endocrine Center, Dallas, Texas
  - Galenos Research, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Spuhler Medical Associates, Friendswood, Texas
  - SMO: Pharmaceuticals C-Trials North Texas Medical Research, Plano, Texas
  - Quality Assurance Research Center Inc, San Antonio, Texas
  - Clinical Trials of Texas Inc, San Antonio, Texas
  - Covenant Clinic Research, San Antonio, Texas
  - Diabetes & Glandular Disease Research Assoc PA, San Antonio, Texas
  - SAM Clinical Research Center, San Antonio, Texas
  - Scott & White Hospital and Clinic, Temple, Texas
  - Pharmaceutical Research Organization, Bountiful, Utah
  - Magna Center for Family Medicine, Magna, Utah
  - Radiant Research Salt Lake City, Salt Lake City, Utah
  - Salt Lake Research, Salt Lake City, Utah
  - Granger Medical Clinic, West Valley City, Utah
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - Sentara Medical Group, Virginia Beach, Virginia
  - Larry D Stonesifer MD Inc PS, Federal Way, Washington
  - Rainier Clinical Research Center Inc, Renton, Washington
  - Cedar Research, Tacoma, Washington
  - Liberty Research Center, Tacoma, Washington
  - Wenatchee Valley Medical Center Clinical Research Department, Wenatchee, Washington
- Brazil (2):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - CPClin-Centro de Pesquisas Clinicas, São Paulo, São Paulo
- Canada (10):
  - Aggarwal and Associates Ltd, Brampton, Ontario
  - Parkwood Hospital, London, Ontario
  - Quest Clinical Trials, Markham, Ontario
  - Lifestyle Metabolism Center, Oakville, Ontario
  - Sarnia Institute of Clinical Research, Sarnia, Ontario
  - The London Road Diagnostic Clinic and Medical Centre, Sarnia, Ontario
  - Lifestyle Metabolism Center, Thornhill, Ontario
  - Lifestyle Metabolism Center, Toronto, Ontario
  - Trial Management Group Inc (Henein, Toronto, Ontario
  - Manna Research, Toronto, Ontario
- Russia (29):
  - Kemerovo State Medical Academy of Ministry of Health, Kemerovo, RUS
  - NHI Kemerovo Regional Clinical Hospital, Kemerovo, RUS
  - NI Principal Military Clinical Hospital n a academician N.N. Burdenko of the Ministry of Defense, Moscow, RUS
  - Moscow State Medical-Stomatological University City Clinical Hospital # 23, Moscow, RUS
  - NEI HPE Moscow State University of Medicine and Dentistry of FAHSD City Clinical Hospital #70, Moscow, RUS
  - Russian State Medical University City Hospital # 4, Moscow, RUS
  - Moscow City Clinical Hospital # 13, Moscow, RUS
  - SHI of Moscow City Clinical Hospital #13, Moscow, RUS
  - NI Central Clinical Hospital of RAS, Moscow, RUS
  - Russian State Medical University Central Clinical Hospital Russian Science Academy, Moscow, RUS
  - City Clinical Hospital # 61, Moscow, RUS
  - SEI HPE Moscow Medical Academy IM Sechenov of Roszdrav Clinic of Endocrinology, Moscow, RUS
  - Russian Scientific Center of Restoration Medicine & Balneology, Moscow, RUS
  - SI Internal Affairs of Moscow- Clinical Hospital, Moscow, RUS
  - RAAMS Endocrinology and Diabetology Department, Moscow, RUS
  - SIH of Moscow City Clinical Hopsital #81 Endocrinology and Diabetology, Moscow, RUS
  - Ryazan State Medical University na academician IP Pavlov, Ryazan, RUS
  - St Petersburg NHI City Polytclinic #77 City Diabetological Center #4, Saint Petersburg, RUS
  - Central Medical Sanitary Unit #122, Saint Petersburg, RUS
  - St Petersburg NHI Municipal Multi-Speciality Hospital # 2, Saint Petersburg, RUS
  - St Petersburg Medical Academy St Elizabeth Hospital, Saint Petersburg, RUS
  - Pavlov State Medical Univ of St Petersburg, Saint Petersburg, RUS
  - TUV Medico-Military Academy, Saint Petersburg, RUS
  - NEI HPE Smolensk State Medical Academy of FAHSD RNHI Smolensk Regional Clinical Hospital, Smolensk, RUS
  - Clinical Pharm Dept of Yaroslavl Clin Hospital, Yaroslavl, RUS
  - MHI Clinical Hospital for Emergency Care na NV Soloviev, Yaroslavl, RUS
  - MCHI Medical Sanitary Unit of Novo-Yaroslavsky Oil Refining Plant, Yaroslavl, RUS
  - NHI Yaroslavl Regional Clinical Hospital, Yaroslavl, RUS
  - Yaroslavl Regional Clinical Hospital, Yaroslavl, RUS